CLINICAL TRIAL: NCT02107001
Title: Lung Ultrasound in Pleuritic Chest Pain: a Multicenter, Prospective, Diagnostic Accuracy Study.
Brief Title: Lung Ultrasound in Pleuritic Chest Pain
Acronym: UPP
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Fabiano Di Marco, M.D., Ph.D., University of Milan
Other Study IDs: UPP08032014
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Community Acquired Pneumonia; Pleuritis; Pulmonary Embolism; Lung Cancer
Keywords: Lung ultrasound; Community acquired p neumonia (CAP); Pleuritis; Pulmonary embolism; Lung Cancer
MeSH Terms: conditions — Community-Acquired Pneumonia; Pleurisy; Pulmonary Embolism; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pleuritic chest pain: Study investigators will perform lung ultrasound in each patient with pleuritic chest pain at inclusion
  Interventions: Procedure: Lung ultrasound

INTERVENTIONS:
Procedure: Lung ultrasound — Lung ultrasonography performed and interpreted by a physician (Pulmonologist or Emergency Physician) possessing specific knowledge in the procedure and a training of at least 100 thoracic ultrasonographies in accordance to a prespecified protocol.
  Other Names: Lung sonography

SUMMARY:
Chest pain is an alarming symptom and one of the most frequent causes of access to the Emergency Departement. Although chest X-ray remains an essential step in the diagnostic process, several studies showed numerous limitations of radiography which frequently is inconclusive. Ultrasonography is a non-radiating imaging technique. Albeit a wide use of ultrasound, the utilization of ultrasound in the study of the lung has only recently been introduced in the clinical practice. Several studies proved that lung ultrasound is useful in the diagnosis of lung consolidation in community acquired pneumonia. Nowadays, ultrasound is not routinely used in the presence of chest pain. Our hypothesis based on clinical experience is that, in patients with pleuritic chest pain, lung ultrasound is very sensitive in detecting pneumonia and other lung diseases (such as pneumothorax) thus performing better than radiography. The primary aim of this study is to verify, in patients affected by pleuritic chest pain, the accuracy of lung ultrasound compared to chest-X-ray. The secondary aim is to evaluate the accuracy of lung ultrasound consolidations in distinguishing lung consolidation in pneumonia, atelectasis, pulmonary infarction, or tumors.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 years and older
* patient affected by thoracic pleuritic pain

Exclusion Criteria:

* patient affected by a chronic condition causing thoracic pain
* patient affected by acute cardiovascular diseases (e.g. acute coronary syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients presenting with pleuritic chest pain referred for medical consultation to italian university and clinical hospitals.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of lung ultrasound in pneumonia, chest wall pain, lung cancer, pulmonary embolism or other causes in patients presenting with pleuritic chest pain. | 30 days
  Sensitivity and specificity, positive and negative predictive values of lung ultrasound in pneumonia, chest wall pain, lung cancer, pulmonary embolism or other causes in patients presenting with pleuritic chest pain.

SECONDARY OUTCOMES:
Accuracy of ultrasound in distinguishing lung consolidation in pneumonia, atelectasis, pulmonary infarction or tumors | 30 days
  Accuracy of ultrasound in differentiating consolidation in distinguishing lung consolidation in pneumonia, atelectasis, pulmonary infarction, tumors or other diseases with respect to the final diagnosis stated by a scientific committee.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Francesco Sferrazza Papa, M.D., Principal Investigator — Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano, Milan, Italy.; Stefano Centanni, M.D, Ph.D., Study Chair — Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano, Milan, Italy.; Giovanni Volpicelli, M.D., Study Director — Emergency Medicine staff Physician San Luigi Gonzaga University Hospital Torino, Italy.
Locations (7):
- Italy (7):
  - Emergency Department, Azienda Ospedaliera Universitaria Careggi, Firenze., Florence
  - USC Pneumologia, Azienda Ospedaliera della Provincia di Lodi, Lodi
  - - U.O.C Broncopneumologia, IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milano., Milan
  - Emergency Department, San Paolo Hospital, Milan
  - Respiratory Unit, San Paolo Hospital, Dipartimento Scienze della Salute, Università degli Studi di Milano., Milan
  - S.O.C. Pneumologia, Ospedale S. Luca, Rovigo., Rovigo
  - - Dipartimento di Medicina d'Urgenza, Ospedale Universitario, S. Luigi Gonzaga, Orbassano (TO)., Turin